CLINICAL TRIAL: NCT06693492
Title: Window On the Brain: Diagnostic, Therapeutic, and Prognostic Sonication of Patients With Disorders of Consciousness
Brief Title: Window On the Brain
Acronym: WOB
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione I.R.C.C.S. Istituto Neurologico Carlo Besta (Other)
Collaborators: IRCCS Istituto delle Scienze Neurologiche di Bologna (Other); S.Anna Rehabilitation Institute (Other); IRCCS Centro Neurolesi Bonino Pulejo (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: PNRR-MAD-2022-12375863
Record Dates: First submitted 2023-12-21; First posted 2024-11-18 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Disorders of Consciousness
Keywords: disorders of consciousness; ultrasound; neuromodulation; minimally conscious state; vegetative state; unresponsive wakefulness syndrome
MeSH Terms: conditions — Consciousness Disorders; Persistent Vegetative State | interventions — Ultrasonography; Diagnosis; Methods

STUDY DESIGN:
Intervention Model Description: Longitudinal prospective cohort study with baseline and follow-up assessment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Chronic patients (DOC duration >=1 year) (Experimental): * Assessment with US technique to characterized the pathophysiological features of chronic DOC
  * For the Interventional part of the project, the selected patients in this arm will be treated with a single session of US neuromodulation and the following measures will be collected before and after the intervention:
  Coma Recovery Scale-revised; Resting state fMRI; EEG-based neurophysiological indices
  Interventions: Device: Ultrasound technique for diagnosis; Focused Ultrasound Stimulation for intervention
- Post-acute patients (DOC duration <1 year) (Experimental): * Assessment with US technique to characterized the pathophysiological features of post-acute DOC and explore its predictive value for chronicization
  * For the Interventional part of the project, the selected patients in this arm will be treated with a single session of US neuromodulation and the following measures will be collected before and after the intervention:
  Coma Recovery Scale-revised; Resting state fMRI; EEG-based neurophysiological indices
  Interventions: Device: Ultrasound technique for diagnosis; Focused Ultrasound Stimulation for intervention

INTERVENTIONS:
Device: Ultrasound technique for diagnosis; Focused Ultrasound Stimulation for intervention — Both chronic and post-acute patients are evaluated through the ultrasound technique to further characterize the mechanisms underlying DOC following acquired brain injuries (e.g., stroke, traumatic brain injury, anoxic events). Furthermore, the predictive value of structural and functional markers for DOC chronicization is explored by following up post-acute DOC patients 1 year after the acute event. Finally, to innovate the therapeutic approach to DOC patients, we adopt the low-intensity focused ultrasound (FUS) on a group of selected 10 patients out of the 100 DOC patients enrolled in the study to modulate brain networks' functioning targeting key brain structures for the recovery of consciousness.

SUMMARY:
Disorders of consciousness (DOC) diagnosis suffers from the difficulty to measure the level of consciousness due to the variability associated with behavioural assessments and the difficulty in detecting the residual level of consciousness in patients who do not show any behavioural signs during the behavioural assessment. This issue could be overcome by using instrumental tools, that are expensive and not always available in clinical settings. The ultrasound-based techniques could represent a valid low-cost and more feasible alternative to deep the knowledge about physio-pathological mechanisms underlying DOC and their chronicization. These techniques could be tailored to treat acute and chronic DOC patients from a personalised medicine perspective. Improving the knowledge, management and care pathways of DOC patients and finding new therapeutic options would benefit not only patients but also public health systems.

DETAILED DESCRIPTION:
After acquired brain injuries, Disorders of Consciousness (DOC) may occur and persist for up to many years. DOC range from Unresponsive Wakefulness Syndrome (UWS; presence of reflexive behaviours) to the emergence from Minimally Conscious State (eMCS; presenting signs of functional communication and/or object use). A correct diagnosis affects the legal decisions, prognosis, and potential therapeutic and rehabilitative interventions. Although DOC diagnosis relies on behavioural assessment (Coma Recovery Scale-Revised; CRS-R), several studies highlight the importance of instrumental tools (e.g., neuroimaging and electrophysiology) for improving diagnosis and prognosis despite their complexity, high costs, and low availability. The ultrasound techniques can represent a valid alternative, allowing both to acquire bedside structural and functional data with low costs and less invasiveness, and perform stimulation to boost consciousness improvement and/or recovery. However, limited evidence exists to date about the use of ultrasound techniques for clinical characterization of DOC patients, and only one registered trial is exploring the effectiveness of ultrasound stimulation for consciousness recovery in this clinical population. For these reasons, we aim to explore the brain functioning and morphology with direct ultrasound (US) in DOC patients, providing both anatomical and functional information in real-time. Specifically, the measures extracted from US examination might provide data regarding DOC's physiopathology in a bedside and affordable manner. Moreover, although clinical trials with low-intensity ultrasound modulation of subcortical structures and thalamic nuclei are already in progress, targeting is still empirical. Thus, understanding US parameters in DOC could provide the ground to improve deep brain structures' targeting, tailoring low-intensity ultrasound parameters according to patient's specific needs for improving their level of consciousness.

ELIGIBILITY:
Aim 1

Inclusion criteria:

* an established diagnosis of DOC (UWS or MCS according to the CRS-R criteria and/or a CRS-R total score ≤22) following severe acquired brain injury;
* age>18 years old;
* written informed consent obtained from each patient's representative.

Exclusion criteria:

* previous psychiatric, neurological, or drug abuse history;
* on-going mechanical ventilation.

From the population enrolled for aim 1, we plan to select ten patients

Inclusion criteria:

* 18<age<65 years;
* medical stability over the previous 30 days;
* presence of the following US variables: low brain stiffness, high elasticity, and adequate level of tissue perfusion;
* written informed consent obtained from each patient's representative;
* structural integrity of both thalami as assessed by MRI.

Exclision criteria:

* contraindications to MRI examination;
* presence of decompressive craniectomy or cranioplasty performed within 30 days;
* presence of epileptogenic features on the EEG and/or drug resistant epileptic crisis history;
* presence of severe muscoloskeletal impairments which are likely to interfere with the correct positioning required for the intervention.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-05-20 (Actual); Primary Completion 2026-05-19 (Estimated); Study Completion 2026-05-19 (Estimated)

PRIMARY OUTCOMES:
Brain ultrasonography measures | T0 (time of enrolment) and T1 (at 6 months from the enrolment for the chronic patients; at 1 year from the acute event for the post-acute patients)
  These data are based on ultrasound parameters extracted from the ultrasound assessment protocol

SECONDARY OUTCOMES:
Level of Consciousness | T0 (time of enrolment) and T1 (at 6 months from the enrolment for the chronic patients; at 1 year from the acute event for the post-acute patients)
  The level of consciousness is derived from the Coma Recovery Scale-revised administration (scale's total score ranges from 0 to 23 where 0 represents the worst clinical condition, fully unconscious, and 23 the best one, fully conscious)
Coma-to-Community outcome measures | T0 (time of enrolment) and T1 (at 6 months from the enrolment for the chronic patients; at 1 year from the acute event for the post-acute patients)
  This measure is represented by the Glasgow Outcome Scale-Extended (GOSE-E), used to measure the clinical outcome after a brain injury. The score ranges from 1 to 8, where 1 represents the worst outcome (i.e. death) and 8 the best possible outcome (i.e. good recovery).
Coma-to-Community outcome measures | T0 (time of enrolment) and T1 (at 6 months from the enrolment for the chronic patients; at 1 year from the acute event for the post-acute patients)
  This measure is represented by the Disability Rating Scale (DRS). The maximum score a patient can obtain on the DRS is 29, which correlates with the vegetative state/unresponsive wakefulness syndrome. A person without disability would score zero.
Neuroendocrine, inflammatory, and nutritional markers derived from a blood sample | T0 (time of enrolment)
  A blood sample will be collected at T0. The rationale is that pituitary dysfunction, chronic inflammation and malnutrition may be associated with a worst outcome and contribute to chronicization.
  The following markers will be collected: haemoglobin, complete blood count, total protein, albumine, transferrine, thyroid stimulating hormone (TSH), free triiodothyronine (FT3), free thyroxine (FT4), cortisol, adrenocorticotropic hormone (ACTH), C-Reactive Protein (PCR), erythrocyte sedimentation rate (ESR), nonfunctioning pituitary tumors (NFT), growth hormone (GH), follicle-stimulating hormone (FSH), luteinizing hormone (LH), prolactin, testosterone and estradiol.
EEG connectivity measures | T0 (time of enrolment)
  Resting state (rs)-EEG will be used to assess and classify patients with DOC. Quantitative EEG measure (Z scored Power Spectral Density, Dominant Frequency peak, and mean Amplitude) wiil be extracted.

CONTACTS AND LOCATIONS:
Locations (4):
- Italy (4):
  - Istituto S. Anna, Semi-Intensive Rehabilitation Unit for Acquired Brain Injury, Crotone, Calabria
  - IRCCS Istituto delle Scienze Neurologiche di Bologna, UO di Medicina Riabilitativa e Neuroriabilitazione, Bologna, Emilia-Romagna
  - Fondazione IRCCS Istituto Neurologico C. Besta, Neurology, Public Helath, Disability Unit, Milan, Lombardy
  - IRCCS Centro Neurolesi Bonino Pulejo, Neuroimaging Lab, Messina, Sicily

IPD SHARING:
Plan to Share IPD: Undecided